CLINICAL TRIAL: NCT01937728
Title: A Randomized, Multicenter, Open Label Study Evaluating the Efficacy and Safety of Tailored Regimens With Peginterferon Alfa-2a Plus Ribavirin According Viral Kinetics for Genotype 1 Chronic Hepatitis C Patients
Brief Title: Tailored Regimens of PEGASYS® and Ribavirin for Genotype 1 Chronic Hepatitis C Patients Trial (TARGET-1)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chia-Yen Dai, Professor, School of Medicine, Hepatology Division, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB-970119
Record Dates: First submitted 2013-06-21; First posted 2013-09-10 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Genotype 1; Peg interferon; alfa 1a; Ribavirin
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A: Peg-interferon alpha-2a & Ribavirin (Active Comparator): Arm A: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 24 weeks with a follow-up period of 24 weeks.
  Interventions: Drug: A: Peg-interferon alpha-2a & Ribavirin
- B: Peg-interferon alpha-2a & Ribavirin (Experimental): Arm B: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 36 weeks with a follow-up period of 24 weeks.
  (Patients who have HVL and an RVR will be randomized into arm B or arm C with a ratio of 1:1)
  Interventions: Drug: B: Peg-interferon alpha-2a & Ribavirin
- C: Peg-interferon alpha-2a & Ribavirin (Experimental): Arm C: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 48 weeks with a follow-up period of 24 weeks.
  (Patients who have HVL and an RVR will be randomized into arm B or arm C with a ratio of 1:1)
  Interventions: Drug: C: Peg-interferon alpha-2a & Ribavirin
- D: Peg-interferon alpha-2a & Ribavirin (Active Comparator): Arm D: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 48 weeks with a follow-up period of 24 weeks.
  (Patients who do not achieve a RVR but have HCV RNA PCR-seronegative at week 12 of treatment)
  Interventions: Drug: D: Peg-interferon alpha-2a & Ribavirin
- E: Peg-interferon alpha-2a & Ribavirin (Experimental): Arm E: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 48 weeks with a follow-up period of 24 weeks.
  (Patients who do not achieve a RVR and remain HCV RNA PCR-seropositive at week 12 of treatment will be randomized into arm E or arm F a ratio of 1:1)
  Interventions: Drug: E: Peg-interferon alpha-2a & Ribavirin
- F: Peg-interferon alpha-2a & Ribavirin (Experimental): Arm F: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 72 weeks with a follow-up period of 24 weeks.
  (Patients who do not achieve a RVR and remain HCV RNA PCR-seropositive at week 12 of treatment will be randomized into arm E or arm F a ratio of 1:1)
  Interventions: Drug: F: Peg-interferon alpha-2a & Ribavirin

INTERVENTIONS:
Drug: A: Peg-interferon alpha-2a & Ribavirin — Arm A: Patients who have low viral loads (LVL, defined as baseline HCV RNA < 400,000 IU/mL) and RVR will be treated with PEGASYS 180ug/week and Ribavirin 1000-1200 mg/day for 24 weeks with a follow-up period of 24 weeks.
  Other Names: Pegasys & Robatrol
  Arms: A: Peg-interferon alpha-2a & Ribavirin
Drug: B: Peg-interferon alpha-2a & Ribavirin — Patients who have HVL and an RVR will be randomized into arm B or arm C with a ratio of 1:1.
  Arm B: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 36 weeks with a follow-up period of 24 weeks.
  Other Names: Pegasys & Robatrol
  Arms: B: Peg-interferon alpha-2a & Ribavirin
Drug: C: Peg-interferon alpha-2a & Ribavirin — Patients who have HVL and an RVR will be randomized into arm B or arm C with a ratio of 1:1.
  Arm C: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 48 weeks with a follow-up period of 24 weeks.
  Other Names: Pegasys, Robatrol
  Arms: C: Peg-interferon alpha-2a & Ribavirin
Drug: D: Peg-interferon alpha-2a & Ribavirin — Arm D: Patients who do not achieve a RVR but have HCV RNA PCR-seronegative at week 12 of treatment will be treated with PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 48 weeks with a follow-up period of 24 weeks.
  Other Names: PEGASYS, Robatrol
  Arms: D: Peg-interferon alpha-2a & Ribavirin
Drug: E: Peg-interferon alpha-2a & Ribavirin — Patients who do not achieve a RVR and remain HCV RNA PCR-seropositive at week 12 of treatment will be randomized into arm E or arm F with a ratio of 1:1.
  Arm E: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 48 weeks with a follow-up period of 24 weeks.
  Other Names: Pegasys, Robatrol
  Arms: E: Peg-interferon alpha-2a & Ribavirin
Drug: F: Peg-interferon alpha-2a & Ribavirin — Patients who do not achieve a RVR and remain HCV RNA PCR-seropositive at week 12 of treatment will be randomized into arm E or arm F with a ratio of 1:1.
  Arm F: PEGASYS® 180 ug/week and Ribavirin 1000-1200 mg/day for 72 weeks with a follow-up period of 24 weeks.
  Other Names: Pegasys, Robatrol
  Arms: F: Peg-interferon alpha-2a & Ribavirin

SUMMARY:
The purposes of this study are:

1. To test if 36 weeks of standard dose of ribavirin with PEGASYS® is non-inferior to standard dose of 48 weeks of ribavirin with PEGASYS® in SVR for patients with RVR and HVL
2. To test if the 72 weeks of treatment with PEGASYS® plus standard dose ribavirin is superior to 48 weeks of the same treatment for patients with HCV RNA seropositivity at week 12

DETAILED DESCRIPTION:
The aims of the present study are:

1. To evaluate the efficacy and safety of 36-week versus 48-week regimen of PEGASYS® (peginterferon alfa-2a, PegIFN) plus standard-dose of ribavirin (RBV) in hepatitis C virus (HCV) genotype 1 infected, treatment-naïve CHC patients who have high viral loads (HVL, defined as baseline HCV RNA ≧ 400,000 IU/mL) and achieve a rapid virologic response (RVR) (defined as seronegativity of HCV RNA at week 4 of treatment)
2. To evaluate the efficacy and safety of 48-week versus 72-week regimen of PegIFN plus standard-dose of RBV in HCV virus genotype 1 infected, treatment-naïve CHC patients with PCR-seropositive of HCV RNA at week 12

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients *18 years of age
* Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribavirin
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Detectable serum HCV-RNA and HCV viral genotype 1
* Liver biopsy findings consistent with the diagnosis of chronic hepatitis C infection with or without compensated cirrhosis (Exception: hemophiliacs in whom biopsy is medically contra-indicated do not require biopsy.)
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using two forms of effective contraception during treatment and during the 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) *6 months prior to the first dose of study drug
* Any investigational drug *6 weeks prior to the first dose of study drug
* Co-infection with active hepatitis A, hepatitis B and/or human immunodeficiency virus (HIV)
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Signs or symptoms of hepatocellular carcinoma
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2010-03; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | 24-week off-treatment period
  Rapid virologic response (RVR), HCV RNA seronegative by PCR at week 4 Sustained virological response (SVR), HCV RNA seronegative by PCR throughout 24-week off-treatment period

SECONDARY OUTCOMES:
Safety | 24-week off-treatment period
  adverse event rate and profile

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yen Dai, M.D., PhD., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan